CLINICAL TRIAL: NCT06510426
Title: Early Interferon-beta Treatment for West-Nile Virus Infection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TLV-0326-24
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: West Nile Virus; West Nile Fever Encephalitis; West Nile Fever Myelitis; West Nile Fever With Other Complications
Keywords: West Nile Virus; WNV; Encephalitis; Flaccid paralysis; WNV neuroinvasive disease
MeSH Terms: conditions — West Nile Fever; Encephalitis | interventions — Interferon beta-1a; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients at high risk for the development of neuroinvasive WNV disease (age 70 and older or immunocompromised patients) or patients presenting with neurologic symptoms of encephalomyelitis will be randomized to receive the study drug or placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): Patients enrolled to participate in the Active Treatment arm will receive 3 subcutaneous injections of 44mcg Interferon b-1a (Rebif), given 48h hours apart.
  Interventions: Drug: Rebif 44 MCG Per 0.5 ML Prefilled Syringe
- Placebo (Placebo Comparator): Patients enrolled to participate in the placebo arm will receive 3 subcutaneous injections of normal saline, given 48h hours apart.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Rebif 44 MCG Per 0.5 ML Prefilled Syringe — Rebif 44mcg per 0.5ml administered subcutaneously
  Arms: Active Treatment
Drug: Saline — 0.5mL of saline administered subcutaneously
  Arms: Placebo

SUMMARY:
West Nile virus (WNV) is a mosquito-borne virus which in majority of cases causes only self-limited disease.

Despite that, in minority of cases (~0.5%) it can infect the brain and cause severe and even life-threatening disease (neuroinvasive disease).

Recent study has shown that up to 40% of WNV patients who develop neuroinvasive disease, have antibodies against Interferons (anti-Type I interferon autoantibodies), which neutralizes interferons, and could explain the development of severe disease.

The investigators therefore assume that early treatment with interferon beta (the type of interferon against which most patients do not have neutralizing antibodies) could prevent the development of severe neuroinvasive WNV disease.

DETAILED DESCRIPTION:
Scientific Background:

West Nile virus (WNV) is a mosquito-borne neurotropic flavivirus that can infect humans and cause life-threatening disease. In recent years, WNV infections have been reported in at least 60 countries across all continents, and is now a leading cause of mosquito-borne disease globally. While most infected individuals remain asymptomatic, around 20% develop a self-limited febrile illness, and less than 1% require hospitalization for neuro-invasive disease. These infrequent, yet severe, neurologic presentations can include encephalitis (50-70%), meningitis (15-35%), and acute flaccid paralysis (3-20%), which can result in a mortality of about 5-20%.

Epidemiologically, age is the strongest known predictor of neuroinvasive disease and death, and the risk of severe disease, particularly neuroinvasive disease, is about 16 times higher in those over the age of 65, and the risk of death is about 30-45 times higher in those over the age of 70.

One possible explanation for the higher risk of older patients to develop more severe disease, is the role of Type I interferons (IFNs) in mediating anti-WNV immunity. In-vitro studies using human cell lines and in-vivo murine models have shown that type-I IFNs can inhibit WNV replication in human cells and protect mice against lethal WNV infection. Even more compelling evidence for the role of type I IFNs in mediating anti-WNV immunity, is a case description of two WNV patients suffering neuroinvasive disease, who improved rapidly after initiation of IFNa treatment.

Accordingly, a recent study has identified very high prevalence of neutralizing anti-Type I IFN autoantibodies in patients with severe WNV neuroinvasive disease. Evaluating nearly 450 patients' samples, anti-Type I IFNs autoantibodies were identified in ~35% of WNV admitted patients and in 40% of those with neuroinvasive disease, including 31% of encephalitis cases, 46% of meningitis cases and 52% of cases of unspecified neurological syndrome. This is in comparison with a prevalence of only 3% in asymptomatic / mild WNV cases.

Of note, the prevalence of neutralizing anti-Type I IFNs auto-antibodies was much higher in patients age 65 and older (45% vs 19%), and to a lesser extent in male patients. In addition, the presence of auto-antibodies neutralizing high concentration of Type-I IFNs (mostly IFNa2) was associated with >100 fold-increase in the risk of neuroinvasive WNV disease, independent of age. These finding suggest that the presence of neutralizing anti-Type I IFN autoantibodies play a role in the development of severe and neuro-invasive WNV disease, and may explain higher risk of severe disease in older individuals.

Regarding the specificity of the anti-Type I IFN autoantibodies; most auto-antibodies were able to neutralize high concentration and super-physiologic concentrations of IFNa2 and /or IFNw(10ng/mL). As for IFNb, no patient had autoantibodies against IFNb only, and only 11% of those having neutralizing antibodies against IFNa2 and/or IFNw also tested positive for neutralizing anti-IFNb autoantibodies, suggesting that IFNb could be potentially used in most patients with WNV disease.

High prevalence of neutralizing anti-Type I IFNs were also identified if patients with severe COVID-19, critical influenza pneumonia and severe adverse reaction to live yellow-fever vaccine.

Based on these finding, a large clinical study showed significant benefit with early administration of a single injection of the Type III IFN, IFN-lambda, in reducing the risk for the development of severe COVID-19 by 50%.

In a similar way, a case report described the use of IFNb in a patient with early COVID-19. The patient, a carrier of an immunodeficiency causing gene, was known to have high concentration of neutralizing anti-Type I IFN auto-antibodies against IFNa and IFNw but no anti-IFNb autoantibodies. A previous patient, carrier of the same immunodeficiency gene, suffered life-threatening COVID-19 pneumonia and displayed neutralizing autoantibodies against type I IFNs.

In an attempt to prevent severe COVID-19, the second patient was treated with 3 doses of IFNb, with rapid resolution of her symptoms.

Taken together, these data suggest the following:

1. Neutralizing anti-Type-I IFN autoantibodies are associated with significantly increased risk for severe and life-threatening viral diseases, including WNV neuroinvasive disease.
2. The prevalence of neutralizing anti-Type-I IFN increases with age, therefore older individuals are at higher risk for developing severe and life-threatening viral diseases.
3. Anti-type I IFN autoantibodies can neutralize high and above physiologic concentrations of type-I IFNs.
4. Most autoantibodies are directed and neutralize IFNa and IFNw and to a lesser extent IFNb
5. Using alternative non-IFNa/w interferons has the potential to bypass this neutralization and prevent progression to severe disease.

For these reasons, the investigators aim to study the protective effect of early IFNb treatment in patients diagnosed with WNV disease.

The rational for using IFNβ is based on the following:

1. Patients with severe or neuroinvasive WNV disease were shown to have high titers of neutralizing autoantibodies against most type I IFNs, including the 13 individual IFNα and IFNω, but less so against IFNβ.
2. The signaling pathway of IFNα and IFNβ is similar, with both binding to the IFNAR1-IFNAR2 heterodimer complex, inducing JAK1/TYK2 activation and STAT1/STAT2 phosphorylation.
3. The known safety profile of subcutaneous injections of IFN-β1a, approved and commonly used for the treatment of relapsing remitting multiple sclerosis.
4. The previously used IFN-lambda is not available in Israel.

Objectives:

Primary objective: To investigate the clinical effects of IFNb1a treatment in patients with a confirmed WNV disease.

Secondary objective: To investigate the prevalence of anti-type-I-IFN autoantibodies in patients with WNV, and their association with clinical outcome of patients with WNV disease.

Research design and methods:

This is a clinical, prospective, double-blinded placebo control trial.

Research process:

1. Patients will be recruited after being diagnosed with WNV either at the ER or after being admitted.
2. Serum, urine and CSF samples from WNV suspected patients will be used to confirm WNV diagnosis based on the presence of either anti-WNV IgM antibodies and/or positive WNV PCR. These samples are collected only for the purpose of establishing a diagnosis, and therefore the volume of the sample collected will be the volume required for establishing a diagnosis (typically 1-2 blood tubes of ~5ml, typical urine sample and 1-2 tubes of CSF samples). Diagnostic studies will be performed at the infectious disease laboratory. Patients will be recruited only after WNV diagnosis is confirmed.
3. Positive patients, if meets inclusion criteria, and after signing an informed consent, will be recruited.
4. Serum and CSF samples from WNV confirmed patients will be collected and stored for later testing for the presence of neutralizing anti-IFN autoantibodies, as well as other potential inflammatory markers. For this purpose, after the establishing of WNV diagnosis, an additional 2 chemistry 6 ml tube (12ml in total) will be collected. CSF samples will not be collected for the purpose of investigational assays, and only if available, residual volumes of CSF collected for the purpose of establishing WNV diagnosis, will be used. These samples will be stored at the Immunology laboratory, and testing for the presence of anti-IFN autoantibodies will be performed at the Clinical Immunology Laboratory.
5. In order to evaluate duration of viremia, blood samples will be collected from the first 30 WNV-confirmed patients, for repeated PCR testing on days 0, day 4 and day 10-14.
6. Patients will be randomized to receive the intervention drug or placebo based on disease manifestation.
7. The intervention drug given will be interferon β1a. Treatment protocol would include 3 subcutaneous injections of IFN-β1a (Rebif), at a dose of 44mcg, given every 48h.
8. Placebo will be normal saline at an equivalent volume to that of the intervention drug, given every 48h.
9. In the case a patient is being discharged before receiving the 3 drug doses, the patient will be invited to receive the remaining doses at the Neurology / Immunology clinic.
10. Patients will be followed for a year after disease onset, with follow-up visits at the neurology clinic every 3 months. Visits would include cognitive and clinical assessments, as well as routine blood work for possible delayed effects of the study drug (including CBC, chemistry with liver and thyroid function) as described in the Schedule of Activities table below .
11. Data regarding 12-month mortality rate will be collected.

Demographics and clinical data will be collected from Chameleon medical record, and will be stored coded on local (TASMC) computers, in a password-protected folder. Folder pathway: W:\West Nile.

No data will be transferred to outside sources.

Randomization process:

Patients will be randomly assigned to each of the two arms with a 1:1 allocation ratio, using randomly selected signed enveloped, considering clinical presentation and neurologic manifestations. For this purpose, stratified block randomization will be implemented, based on the 3 possible strata generated from the two binary variables (presence or absence of neurologic symptoms; in case of neurologic symptoms, presence or absence of flaccid paralysis). A randomization code will be given and maintained for the duration of the study. A planned breaking of randomization codes will be performed and reviewed by an independent Data and Safety Monitoring Board as explained below. There will be no planned breaking by the blinded researchers . Unplanned breaking of codes to team or patient would lead to exclusion of the patient from the analysis.

The study drug and placebo will be prepared in the clinical research unit, at the pharmacy of the Tel-Aviv Sourasky Medical Center, by a certified pharmacist, in accordance with procedure #135 of the Pharmaceutics Division (Ministry of Health).

The study drug / placebo will be labeled with the following: study title; protocol number; name of PI; name of study drug / placebo (both); randomization number; date and time of preparation;

ELIGIBILITY:
Diagnosis of WNV infection will be based on the following:

1. Patients with clinical presentation suspected as compatible with WNV infection, with symptoms including elevated fever, headache or flaccid paralysis or fever with encephalopathy.

   And:
2. Positive anti-WNV IgM serology / WNV PCR from either serum, urine or CSF.

Inclusion criteria:

We aim to focus on three patients' populations:

1. Patients older than 70 years of age, who are at higher risk for the presence of neutralizing anti-Type I IFN auto-antibodies, and therefore at higher risk for developing severe neuroinvasive disease. Only patients who fulfill the diagnostic criteria above will be included.
2. Patients presenting with neuroinvasive WNV disease, including either flaccid paralysis or encephalitis, independent of their age, excluding a presentation consistent with isolated aseptic meningitis (headache, fever, 6th nerve palsy). Only patients who fulfill the diagnostic criteria above will be included.
3. Immunocompromised patients at any age. Immunocompromised patients will be defined as patients with hematologic malignancy (treated or untreated); chemotherapy within previous 4 weeks, stem cell transplant recipient or solid organ transplant recipient; use of any immunosuppressant drug including prednisone greater than or equal to 20 mg/day within the previous 4 weeks; primary / acquired immunodeficiency disorder. Only patients who fulfill the diagnostic criteria above will be included.

Exclusion Criteria:

1. Patients younger than 18 years old.
2. Pregnant women.
3. Contraindication for the administration of the drug: Hypersensitivity to natural or recombinant interferon beta, and decompensated liver disease.
4. A patient with neuroinvasive disease showing consistent spontaneous improvement over a period of > 2 days and mRS of below 4.
5. More than 8 days from onset of neurological symptoms in immunocompetent patients and more than 10 days in immunocompromised patients. This time frame will be renewed if a patient with flaccid paralysis develops new onset encephalitis.
6. Patients who are receiving active chemotherapy treatment or suffer concurrent severe viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of death or intubation | 4 weeks
  Death or intubation within 4 weeks
Modified Rankin Scale (mRS) score | 3 and 6 months
  Comparison of modified Rankin Scale (mRS) score at 3 and 6 months. The mRS score is a 7 point (0-6) disability scale with higher score suggesting higher level of disability.

SECONDARY OUTCOMES:
ICU admission | 4 weeks
  Rates of ICU admission
Mechanical ventilation | 4 weeks
  Rates of mechanical ventilation
Modified-NIH-stroke-scale (mNIHSS) | 3 months
  Change in modified-NIH-stroke-scale (mNIHSS) from baseline to 3 months. The scoring range is 0 to 42 points, with higher numbers indicating greater severity.
Mini-mental state examination (MMSE) | 3 months
  Change in mini-mental state examination (MMSE) from baseline to 3 months. The MMSE has a range score of 0-30. A higher score suggests better performance. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
All cause mortality | 12 months
  All-cause mortality at 4 weeks, 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Gervais A, Rovida F, Avanzini MA, Croce S, Marchal A, Lin SC, Ferrari A, Thorball CW, Constant O, Le Voyer T, Philippot Q, Rosain J, Angelini M, Perez Lorenzo M, Bizien L, Achille C, Trespidi F, Burdino E, Cassaniti I, Lilleri D, Fornara C, Sammartino JC, Cereda D, Marrocu C, Piralla A, Valsecchi C, Ricagno S, Cogo P, Neth O, Marin-Cruz I, Pacenti M, Sinigaglia A, Trevisan M, Volpe A, Marzollo A, Conti F, Lazzarotto T, Pession A, Viale P, Fellay J, Ghirardello S, Aubart M, Ghisetti V, Aiuti A, Jouanguy E, Bastard P, Percivalle E, Baldanti F, Puel A, MacDonald MR, Rice CM, Rossini G, Murray KO, Simonin Y, Nagy A, Barzon L, Abel L, Diamond MS, Cobat A, Zhang SY, Casanova JL, Borghesi A. Autoantibodies neutralizing type I IFNs underlie West Nile virus encephalitis in approximately 40% of patients. J Exp Med. 2023 Sep 4;220(9):e20230661. doi: 10.1084/jem.20230661. Epub 2023 Jun 22. PMID 37347462
- [Background] Schoggins JW, Wilson SJ, Panis M, Murphy MY, Jones CT, Bieniasz P, Rice CM. A diverse range of gene products are effectors of the type I interferon antiviral response. Nature. 2011 Apr 28;472(7344):481-5. doi: 10.1038/nature09907. Epub 2011 Apr 10. PMID 21478870
- [Background] Samuel MA, Diamond MS. Alpha/beta interferon protects against lethal West Nile virus infection by restricting cellular tropism and enhancing neuronal survival. J Virol. 2005 Nov;79(21):13350-61. doi: 10.1128/JVI.79.21.13350-13361.2005. PMID 16227257
- [Background] Bastard P, Rosen LB, Zhang Q, Michailidis E, Hoffmann HH, Zhang Y, Dorgham K, Philippot Q, Rosain J, Beziat V, Manry J, Shaw E, Haljasmagi L, Peterson P, Lorenzo L, Bizien L, Trouillet-Assant S, Dobbs K, de Jesus AA, Belot A, Kallaste A, Catherinot E, Tandjaoui-Lambiotte Y, Le Pen J, Kerner G, Bigio B, Seeleuthner Y, Yang R, Bolze A, Spaan AN, Delmonte OM, Abers MS, Aiuti A, Casari G, Lampasona V, Piemonti L, Ciceri F, Bilguvar K, Lifton RP, Vasse M, Smadja DM, Migaud M, Hadjadj J, Terrier B, Duffy D, Quintana-Murci L, van de Beek D, Roussel L, Vinh DC, Tangye SG, Haerynck F, Dalmau D, Martinez-Picado J, Brodin P, Nussenzweig MC, Boisson-Dupuis S, Rodriguez-Gallego C, Vogt G, Mogensen TH, Oler AJ, Gu J, Burbelo PD, Cohen JI, Biondi A, Bettini LR, D'Angio M, Bonfanti P, Rossignol P, Mayaux J, Rieux-Laucat F, Husebye ES, Fusco F, Ursini MV, Imberti L, Sottini A, Paghera S, Quiros-Roldan E, Rossi C, Castagnoli R, Montagna D, Licari A, Marseglia GL, Duval X, Ghosn J; HGID Lab; NIAID-USUHS Immune Response to COVID Group; COVID Clinicians; COVID-STORM Clinicians; Imagine COVID Group; French COVID Cohort Study Group; Milieu Interieur Consortium; CoV-Contact Cohort; Amsterdam UMC Covid-19 Biobank; COVID Human Genetic Effort; Tsang JS, Goldbach-Mansky R, Kisand K, Lionakis MS, Puel A, Zhang SY, Holland SM, Gorochov G, Jouanguy E, Rice CM, Cobat A, Notarangelo LD, Abel L, Su HC, Casanova JL. Autoantibodies against type I IFNs in patients with life-threatening COVID-19. Science. 2020 Oct 23;370(6515):eabd4585. doi: 10.1126/science.abd4585. Epub 2020 Sep 24. PMID 32972996
- [Background] Bastard P, Gervais A, Le Voyer T, Rosain J, Philippot Q, Manry J, Michailidis E, Hoffmann HH, Eto S, Garcia-Prat M, Bizien L, Parra-Martinez A, Yang R, Haljasmagi L, Migaud M, Sarekannu K, Maslovskaja J, de Prost N, Tandjaoui-Lambiotte Y, Luyt CE, Amador-Borrero B, Gaudet A, Poissy J, Morel P, Richard P, Cognasse F, Troya J, Trouillet-Assant S, Belot A, Saker K, Garcon P, Riviere JG, Lagier JC, Gentile S, Rosen LB, Shaw E, Morio T, Tanaka J, Dalmau D, Tharaux PL, Sene D, Stepanian A, Megarbane B, Triantafyllia V, Fekkar A, Heath JR, Franco JL, Anaya JM, Sole-Violan J, Imberti L, Biondi A, Bonfanti P, Castagnoli R, Delmonte OM, Zhang Y, Snow AL, Holland SM, Biggs C, Moncada-Velez M, Arias AA, Lorenzo L, Boucherit S, Coulibaly B, Anglicheau D, Planas AM, Haerynck F, Duvlis S, Nussbaum RL, Ozcelik T, Keles S, Bousfiha AA, El Bakkouri J, Ramirez-Santana C, Paul S, Pan-Hammarstrom Q, Hammarstrom L, Dupont A, Kurolap A, Metz CN, Aiuti A, Casari G, Lampasona V, Ciceri F, Barreiros LA, Dominguez-Garrido E, Vidigal M, Zatz M, van de Beek D, Sahanic S, Tancevski I, Stepanovskyy Y, Boyarchuk O, Nukui Y, Tsumura M, Vidaur L, Tangye SG, Burrel S, Duffy D, Quintana-Murci L, Klocperk A, Kann NY, Shcherbina A, Lau YL, Leung D, Coulongeat M, Marlet J, Koning R, Reyes LF, Chauvineau-Grenier A, Venet F, Monneret G, Nussenzweig MC, Arrestier R, Boudhabhay I, Baris-Feldman H, Hagin D, Wauters J, Meyts I, Dyer AH, Kennelly SP, Bourke NM, Halwani R, Sharif-Askari NS, Dorgham K, Sallette J, Sedkaoui SM, AlKhater S, Rigo-Bonnin R, Morandeira F, Roussel L, Vinh DC, Ostrowski SR, Condino-Neto A, Prando C, Bonradenko A, Spaan AN, Gilardin L, Fellay J, Lyonnet S, Bilguvar K, Lifton RP, Mane S; HGID Lab; COVID Clinicians; COVID-STORM Clinicians; NIAID Immune Response to COVID Group; NH-COVAIR Study Group; Danish CHGE; Danish Blood Donor Study; St. James's Hospital; SARS CoV2 Interest group; French COVID Cohort Study Group; Imagine COVID-Group; Milieu Interieur Consortium; CoV-Contact Cohort; Amsterdam UMC Covid-19; Biobank Investigators; COVID Human Genetic Effort; CONSTANCES cohort; 3C-Dijon Study; Cerba Health-Care; Etablissement du Sang study group; Anderson MS, Boisson B, Beziat V, Zhang SY, Vandreakos E, Hermine O, Pujol A, Peterson P, Mogensen TH, Rowen L, Mond J, Debette S, de Lamballerie X, Duval X, Mentre F, Zins M, Soler-Palacin P, Colobran R, Gorochov G, Solanich X, Susen S, Martinez-Picado J, Raoult D, Vasse M, Gregersen PK, Piemonti L, Rodriguez-Gallego C, Notarangelo LD, Su HC, Kisand K, Okada S, Puel A, Jouanguy E, Rice CM, Tiberghien P, Zhang Q, Cobat A, Abel L, Casanova JL. Autoantibodies neutralizing type I IFNs are present in ~4% of uninfected individuals over 70 years old and account for ~20% of COVID-19 deaths. Sci Immunol. 2021 Aug 19;6(62):eabl4340. doi: 10.1126/sciimmunol.abl4340. PMID 34413139
- [Background] Zhang Q, Pizzorno A, Miorin L, Bastard P, Gervais A, Le Voyer T, Bizien L, Manry J, Rosain J, Philippot Q, Goavec K, Padey B, Cupic A, Laurent E, Saker K, Vanker M, Sarekannu K; COVID Human Genetic Effort; Etablissement Francais du Sang Study Group; Constances Cohort; 3C-Dijon Study; Cerba HealthCare Group; Lyon Antigrippe Working Group; REIPI INF Working Group; Garcia-Salum T, Ferres M, Le Corre N, Sanchez-Cespedes J, Balsera-Manzanero M, Carratala J, Retamar-Gentil P, Abelenda-Alonso G, Valiente A, Tiberghien P, Zins M, Debette S, Meyts I, Haerynck F, Castagnoli R, Notarangelo LD, Gonzalez-Granado LI, Dominguez-Pinilla N, Andreakos E, Triantafyllia V, Rodriguez-Gallego C, Sole-Violan J, Ruiz-Hernandez JJ, Rodriguez de Castro F, Ferreres J, Briones M, Wauters J, Vanderbeke L, Feys S, Kuo CY, Lei WT, Ku CL, Tal G, Etzioni A, Hanna S, Fournet T, Casalegno JS, Queromes G, Argaud L, Javouhey E, Rosa-Calatrava M, Cordero E, Aydillo T, Medina RA, Kisand K, Puel A, Jouanguy E, Abel L, Cobat A, Trouillet-Assant S, Garcia-Sastre A, Casanova JL. Autoantibodies against type I IFNs in patients with critical influenza pneumonia. J Exp Med. 2022 Nov 7;219(11):e20220514. doi: 10.1084/jem.20220514. Epub 2022 Sep 16. PMID 36112363
- [Background] Bastard P, Michailidis E, Hoffmann HH, Chbihi M, Le Voyer T, Rosain J, Philippot Q, Seeleuthner Y, Gervais A, Materna M, de Oliveira PMN, Maia MLS, Dinis Ano Bom AP, Azamor T, Araujo da Conceicao D, Goudouris E, Homma A, Slesak G, Schafer J, Pulendran B, Miller JD, Huits R, Yang R, Rosen LB, Bizien L, Lorenzo L, Chrabieh M, Erazo LV, Rozenberg F, Jeljeli MM, Beziat V, Holland SM, Cobat A, Notarangelo LD, Su HC, Ahmed R, Puel A, Zhang SY, Abel L, Seligman SJ, Zhang Q, MacDonald MR, Jouanguy E, Rice CM, Casanova JL. Auto-antibodies to type I IFNs can underlie adverse reactions to yellow fever live attenuated vaccine. J Exp Med. 2021 Apr 5;218(4):e20202486. doi: 10.1084/jem.20202486. PMID 33544838
- [Background] de Weerd NA, Vivian JP, Nguyen TK, Mangan NE, Gould JA, Braniff SJ, Zaker-Tabrizi L, Fung KY, Forster SC, Beddoe T, Reid HH, Rossjohn J, Hertzog PJ. Structural basis of a unique interferon-beta signaling axis mediated via the receptor IFNAR1. Nat Immunol. 2013 Sep;14(9):901-7. doi: 10.1038/ni.2667. Epub 2013 Jul 21. PMID 23872679
- [Result] Kalil AC, Devetten MP, Singh S, Lesiak B, Poage DP, Bargenquast K, Fayad P, Freifeld AG. Use of interferon-alpha in patients with West Nile encephalitis: report of 2 cases. Clin Infect Dis. 2005 Mar 1;40(5):764-6. doi: 10.1086/427945. Epub 2005 Feb 7. PMID 15714427
- [Result] Reis G, Moreira Silva EAS, Medeiros Silva DC, Thabane L, Campos VHS, Ferreira TS, Santos CVQ, Nogueira AMR, Almeida APFG, Savassi LCM, Figueiredo-Neto AD, Dias ACF, Freire Junior AM, Bitaraes C, Milagres AC, Callegari ED, Simplicio MIC, Ribeiro LB, Oliveira R, Harari O, Wilson LA, Forrest JI, Ruton H, Sprague S, McKay P, Guo CM, Limbrick-Oldfield EH, Kanters S, Guyatt GH, Rayner CR, Kandel C, Biondi MJ, Kozak R, Hansen B, Zahoor MA, Arora P, Hislop C, Choong I, Feld JJ, Mills EJ, Glenn JS; TOGETHER Investigators. Early Treatment with Pegylated Interferon Lambda for Covid-19. N Engl J Med. 2023 Feb 9;388(6):518-528. doi: 10.1056/NEJMoa2209760. PMID 36780676
- [Result] Bastard P, Levy R, Henriquez S, Bodemer C, Szwebel TA, Casanova JL. Interferon-beta Therapy in a Patient with Incontinentia Pigmenti and Autoantibodies against Type I IFNs Infected with SARS-CoV-2. J Clin Immunol. 2021 Jul;41(5):931-933. doi: 10.1007/s10875-021-01023-5. Epub 2021 Mar 25. No abstract available. PMID 33763778